CLINICAL TRIAL: NCT05006885
Title: A Phase 1, 12-Week, Randomized, Double-Blind, Placebo-Controlled Study of ALT-801 in Diabetic and Non-Diabetic Overweight and Obese Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: ALT-801 in Diabetic and Non-Diabetic Overweight and Obese Subjects With Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-801-105
Record Dates: First submitted 2021-07-30; First posted 2021-08-16 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Obese; Overweight
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Overweight | interventions — ALT-801

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ALT-801 Dose Level 1 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 2 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- ALT-801 Dose Level 3 (Experimental): Administered once a week for 12 weeks
  Interventions: Drug: ALT-801
- Placebo (Placebo Comparator): Administered once a week for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALT-801 — Injected subcutaneously (SC)
  Other Names: Pemvidutide
  Arms: ALT-801 Dose Level 1; ALT-801 Dose Level 2; ALT-801 Dose Level 3
Other: Placebo — Injected subcutaneously (SC)
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety and tolerability of ALT-801 in diabetic and non-diabetic subjects with overweight and obese and non-alcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, randomized, double-blind, placebo-controlled study to assess the effects of ALT-801 the safety of ALT-801and effects on hepatic fat fraction, anthropometric parameters, lipid metabolism, inflammatory markers and fibrosis markers in diabetic and non-diabetic overweight and obese (BMI 28.0-45.0 kg/m2) subjects with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed prior to the performance of any study procedures
* Male or female volunteers, age 18 to 65 years, inclusive
* Overweight to obese (greater than or equal to BMI 28.0
* Magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) ≥ 10%
* If subject has Type 2 diabetes mellitus (T2DM), on stable regimen, for at least 3 months prior to screening, of any combination (1) diet and exercise, (2) metformin with absent or mild gastrointestinal symptoms (nausea, vomiting or diarrhea), and/or (3) sodium glucose cotransporter-2 (SGLT-2) therapy

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Type 1 DM and/or insulin-dependent T2DM, or uncontrolled T2DM defined as HbA1c ≥ 9.5%
* History of pancreatitis or hypersensitivity reaction to GLP-1 analogues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
The Number of Participants with One or More Treatment-Emergent Adverse Events (TEAEs) | Up to Day 110
  Number of participants with 1 or more TEAEs up to Day 110

SECONDARY OUTCOMES:
Change from baseline in liver fat fraction by MRI-PDFF | Baseline and Day 85
  Change in liver fat fraction by MRI-PDFF from Baseline to Day 85
Change from baseline in body weight | Baseline and Day 85
  Change in body weight from Baseline to Day 85
Change from baseline in lipid metabolism (total cholesterol, HDL cholesterol, LDL cholesterol, lipoprotein fractions) | Baseline and Day 85
  Change from in lipid metabolism (TC, HDL, LDL) from Baseline to Day 85
Change from baseline in hemoglobin A1c | Baseline and Day 85
  Change in hemoglobin A1c from Baseline to Day 85
Change from baseline in fibrosis markers (Pro-C3) | Baseline and Day 85
  Change in fibrosis markers (Pro-C3) from Baseline to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Browne, MD, Study Director — Altimmune, Inc.
Locations (15):
- United States (15):
  - Headlands Research Scottsdale, Scottsdale, Arizona
  - QLMC, Tucson, Arizona
  - Catalina Research Institute, Montclair, California
  - Clinical Trials Research, Sacramento, California
  - Panax Clinical Research, Miami Lakes, Florida
  - Covenant Research and Clinics, Sarasota, Florida
  - Headlands Research Sarasota, Sarasota, Florida
  - Wake Research CRCN, Las Vegas, Nevada
  - Accelemed Research Institute, Austin, Texas
  - Pinnacle Research, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Pinnacle Research, San Antonio, Texas
  - Cognitive Clinical Trials, Salt Lake City, Utah

REFERENCES:
- [Derived] Harrison SA, Browne SK, Suschak JJ, Tomah S, Gutierrez JA, Yang J, Roberts MS, Harris MS. Effect of pemvidutide, a GLP-1/glucagon dual receptor agonist, on MASLD: A randomized, double-blind, placebo-controlled study. J Hepatol. 2025 Jan;82(1):7-17. doi: 10.1016/j.jhep.2024.07.006. Epub 2024 Jul 11. PMID 39002641